CLINICAL TRIAL: NCT03772626
Title: The Feasibility and Efficacy of Heated Humidified Nasal Cannula (AIRVOTM) in Hospital and at Home - An Open-Label, Non-Randomized Pilot Study.
Brief Title: Heated High Humidity After COPD Exacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Joshua Wald, Assistant Professor Department of Medicine, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Heated Humidity after COPDE
Record Dates: First submitted 2018-12-06; First posted 2018-12-11 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: COPD Exacerbation
Keywords: COPD; Heated humidified high-flow nasal cannula; Exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Single group non-randomized open label study of efficacy and feasibility. Comparison will be to historical controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Heated humidified high-flow (Experimental): Heated Humidified High-flow Nasal Cannula
  Interventions: Device: Heated Humidified High-flow Nasal Cannula

INTERVENTIONS:
Device: Heated Humidified High-flow Nasal Cannula — Patients will receive heated high humidity air through the AIRVO(TM) device starting in hospital and continuing for 60 days after hospital discharge. Oxygen will be titrated to target SpO2 between 88-92%, patients not requiring oxygen will receive heated high humidity air without oxygen. Temperature and flow rate will titrated to patient comfort with a target temperature 37 degree Celsius and flow rate of ≥20 l/minute. Patients will be encouraged to use the device overnight and when needed during the day with a target duration of at least 6 hours per night

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease usually caused by exposure to tobacco smoke which leads to chronic symptoms of shortness of breath, cough, and phlegm. COPD is one of the leading causes of disability and death in Canada. Individuals with COPD often have periodic worsening of their disease, called exacerbations, consisting of increased shortness of breath and often an increase in cough and phlegm. These exacerbations often lead to hospital admission and are associated with worsening symptoms and lung function over time. After an exacerbation individuals with COPD usually take several weeks to return to their previous state of health and many people with an exacerbation who are discharged from hospital return to the ER within 60. Heated humidified air has been shown to improve the clearance of mucous in the lungs for people with chronic lung disease. By providing patients at St. Joseph's Hospital who are discharged after a COPD exacerbation with a device for delivering heated high humidity air to use overnight it is hoped that these individuals will be able to more easily keep their lungs and airways free of mucous. This in turn may lead to improvement in their symptoms of shortness of breath, cough, and phlegm production as well as decreasing obstruction of the airways to reduce the risk of having to return to the emergency room or hospital.

DETAILED DESCRIPTION:
COPD is a respiratory condition that is often associated with cigarette smoking, and defined by incompletely reversible airflow obstruction and complicated by exacerbations. Mucous hypersecretion with impaired mucociliary transport are frequently present, and are associated with infective AECOPD, and death related to pulmonary infection. COPD is both common, affecting 1 in 6 Canadians, and burdensome, being the 4th leading cause of death, in the Canadian population.

In Canada, the most common primary diagnosis associated with admission to hospital is acute exacerbation of COPD (AECOPD). For moderate to severe COPD, the average patient will have more than 2 AECOPD per year. A single episode conveys a poor prognosis, being associated with death, further AECOPD events, and reduced health-related quality of life. Despite multiple guideline-based management strategies, 1 in 3 patients with AECOPD will have another episode within 8 weeks.

Although the technology for heated humidified high-flow nasal cannula (HFNC) has been available for two decades, it has only recently become widely available for adults. The rapid humidification of gas allows this system to achieve flow rates of up to 60 liters per minute. These two factors, in combination, allow for a higher achieved fraction of inspired oxygen, and benefit the expectoration of secretions and ventilatory efficiency. Randomised clinical trials of ICU patients have demonstrated that HFNC is non-inferior to non-invasive ventilation both in the setting of acute hypoxemic respiratory failure and as an adjunct therapy post-extubation.

HFNC is a promising treatment for patients with COPD as it can counteract potentially harmful mucous abnormalities by reducing mucous viscosity and restoring mucociliary transport. Randomised studies have also demonstrated that HFNC administered at home results in an increased the time to first exacerbation, fewer AECOPD, improved quality-of-life, and reduced PaCO2. However, the efficacy of HFNC during hospital admission, when mucous abnormalities and poor expectoration could be most pronounced, has not yet been studied. Furthermore, the feasibility and efficacy of this device as a patient transitions from the hospital to the community after an AECOPD remains to be elucidated.

The objectives of this study are to test the efficacy of a heated humidified high-flow nasal cannula used during and after a hospital admission for AECOPD to reduce the risk of return to ER or readmission, and the feasibility of implementing such a device starting in hospital with transition to the home environment.

This is an open-label, non-randomized pilot study of in-hospital and home HFNC in patients with COPD. Patients who consent to participate will have an a heated humidified high-flow nasal cannula device configured by a respiratory therapist and available at their bedside in hospital. Fraction of inspired oxygen will be adjusted as needed to obtain a pulse oximetry reading between 88-92%. If hypoxemia is not present (peripheral oxygen saturation (SpO2) ≥88%) on room air, then the device will be used without supplemental oxygen. Temperature and flow rate will be titrated for patient comfort with a target temperature of 37 degrees Celsius and flow rate of ≥20 liters per minute if tolerated. Participants will be instructed to use the device overnight and as much as they like during the day targeting at least 6 hours of use per 24 hour period.

At discharge, subjects will be provided with a heated humidified high-flow nasal cannula home device. Targeted use and oxygen titration will remain unchanged from inpatient use. A respiratory therapist from will perform a home visit within 24 hours of hospital discharge to educate the patient on home use and ensure proper set up of the device, and an additional visit 2 weeks post-discharge. Patients will have access to a 24 hour emergency telephone number if they have any concerns. The duration of the trial will be 60 days post-discharge after which the device will be returned.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Hospital with a primary diagnosis of exacerbation of COPD
* Greater then or equal to 20 pack year history of smoking
* Participating in Integrated Comprehensive Care (ICC) home care program

Exclusion Criteria:

* Requirement for acute non-invasive ventilation in hospital
* Use of nocturnal non-invasive ventilation prior to hospitalization

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
ER use or hospitalization for COPD | Length of study participation (60 days after hospital discharge)
  ER visits or hospital admissions for COPD during the 60 day treatment period

SECONDARY OUTCOMES:
Hospital length of stay | Collected throughout inpatient enrollment period until last enrolled patient discharged (Expected total of 70 days)
  Total length of stay in hospital during index admission for COPD
Use of home-care resources | Length of study participation (60 days after hospital discharge)
  Total number of unplanned home visits during study period

OTHER OUTCOMES:
Average daily use of heated humidified high-flow nasal cannula | Length of study participation (60 days after hospital discharge)
  number of hours of machine use divided by days enrolled in study
Number of eligible patients who consent to the trial | Collected throughout inpatient enrollment period (total of 60 days)
  Proportion of eligible patients who consent will be calculated
Drop out rate | Length of study participation (60 days after hospital discharge)
  Proportion of patients who enroll in the trial who successfully complete the trial
Patient satisfaction with heated humidified high-flow nasal cannula | Collected at end of study participartion (60 days after hospital discharge)
  brief survey created for the study to measure patient satisfaction with the device. 5 questions, each individual item will be rated on a 5 part Likert scale from 1 = strongly agree to 5 = strongly disagree with a 1 indicating the highest satisfaction and a 5 indicating the lowest satisfaction. Results for each question will be reported separately.
Nursing satisfaction with heated humidified high-flow nasal cannula in hospital | Collected throughout inpatient enrollment period (total of 60 days)
  Anonymous satisfaction survey given to nurses on medical units, brief survey created for the study to measure nursing satisfaction with the device. 5 questions, each individual item will be rated on a 5 part Likert scale from 1 = strongly agree to 5 = strongly disagree with a 1 indicating the highest satisfaction and a 5 indicating the lowest satisfaction. Results for each question will be reported separately.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wald, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Donnell DE, Aaron S, Bourbeau J, Hernandez P, Marciniuk DD, Balter M, Ford G, Gervais A, Goldstein R, Hodder R, Kaplan A, Keenan S, Lacasse Y, Maltais F, Road J, Rocker G, Sin D, Sinuff T, Voduc N. Canadian Thoracic Society recommendations for management of chronic obstructive pulmonary disease - 2007 update. Can Respir J. 2007 Sep;14 Suppl B(Suppl B):5B-32B. doi: 10.1155/2007/830570. PMID 17885691
- [Background] Rogers DF. The role of airway secretions in COPD: pathophysiology, epidemiology and pharmacotherapeutic options. COPD. 2005 Sep;2(3):341-53. doi: 10.1080/15412550500218098. PMID 17146999
- [Background] Prescott E, Lange P, Vestbo J. Chronic mucus hypersecretion in COPD and death from pulmonary infection. Eur Respir J. 1995 Aug;8(8):1333-8. doi: 10.1183/09031936.95.08081333. PMID 7489800
- [Background] Gershon AS, Thiruchelvam D, Chapman KR, Aaron SD, Stanbrook MB, Bourbeau J, Tan W, To T; Canadian Respiratory Research Network. Health Services Burden of Undiagnosed and Overdiagnosed COPD. Chest. 2018 Jun;153(6):1336-1346. doi: 10.1016/j.chest.2018.01.038. Epub 2018 Feb 6. PMID 29425675
- [Background] O'Donnell DE, Hernandez P, Kaplan A, Aaron S, Bourbeau J, Marciniuk D, Balter M, Ford G, Gervais A, Lacasse Y, Maltais F, Road J, Rocker G, Sin D, Sinuff T, Voduc N. Canadian Thoracic Society recommendations for management of chronic obstructive pulmonary disease - 2008 update - highlights for primary care. Can Respir J. 2008 Jan-Feb;15 Suppl A(Suppl A):1A-8A. doi: 10.1155/2008/641965. PMID 18292855
- [Background] Keene JD, Jacobson S, Kechris K, Kinney GL, Foreman MG, Doerschuk CM, Make BJ, Curtis JL, Rennard SI, Barr RG, Bleecker ER, Kanner RE, Kleerup EC, Hansel NN, Woodruff PG, Han MK, Paine R 3rd, Martinez FJ, Bowler RP, O'Neal WK; COPDGene and SPIROMICS Investigators double dagger. Biomarkers Predictive of Exacerbations in the SPIROMICS and COPDGene Cohorts. Am J Respir Crit Care Med. 2017 Feb 15;195(4):473-481. doi: 10.1164/rccm.201607-1330OC. PMID 27579823
- [Background] Connors AF Jr, Dawson NV, Thomas C, Harrell FE Jr, Desbiens N, Fulkerson WJ, Kussin P, Bellamy P, Goldman L, Knaus WA. Outcomes following acute exacerbation of severe chronic obstructive lung disease. The SUPPORT investigators (Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments). Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):959-67. doi: 10.1164/ajrccm.154.4.8887592.
- [Background] Groenewegen KH, Schols AM, Wouters EF. Mortality and mortality-related factors after hospitalization for acute exacerbation of COPD. Chest. 2003 Aug;124(2):459-67. doi: 10.1378/chest.124.2.459. PMID 12907529
- [Background] Pradan L, Ferreira I, Postolache P. The quality of medical care during an acute exacerbations of chronic obstructive pulmonary disease. Rev Med Chir Soc Med Nat Iasi. 2013 Oct-Dec;117(4):870-4. PMID 24502063
- [Background] Donaldson GC, Wedzicha JA. COPD exacerbations .1: Epidemiology. Thorax. 2006 Feb;61(2):164-8. doi: 10.1136/thx.2005.041806. PMID 16443707
- [Background] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Background] Rea H, McAuley S, Jayaram L, Garrett J, Hockey H, Storey L, O'Donnell G, Haru L, Payton M, O'Donnell K. The clinical utility of long-term humidification therapy in chronic airway disease. Respir Med. 2010 Apr;104(4):525-33. doi: 10.1016/j.rmed.2009.12.016. Epub 2010 Feb 9. PMID 20144858
- [Background] Storgaard LH, Hockey HU, Laursen BS, Weinreich UM. Long-term effects of oxygen-enriched high-flow nasal cannula treatment in COPD patients with chronic hypoxemic respiratory failure. Int J Chron Obstruct Pulmon Dis. 2018 Apr 16;13:1195-1205. doi: 10.2147/COPD.S159666. eCollection 2018. PMID 29713153